CLINICAL TRIAL: NCT07254039
Title: Development and Validation of an AI-Assisted Electrochemical Sensor Platform for Saliva-Based Diagnostics in Periodontitis
Brief Title: AI-Assisted Saliva Diagnostics Using an Electrochemical Sensor Platform for Periodontitis Detection (SALIENCE)
Acronym: SALIENCE
Status: Not yet recruiting | Type: Observational
Sponsor: Ostergotland County Council, Sweden (Other)
Collaborators: Malmö University (Other); Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Shariel Sayardoust, Associate Professor, Ostergotland County Council, Sweden
Other Study IDs: SALIENCE2025
Record Dates: First submitted 2025-11-15; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Periodontal Diseases; Biomarkers (D23.050.301); Diagnostic; Saliva
Keywords: Saliva Diagnostics; Electrochemical Sensor; AI-Assisted Diagnostics; Biomarkers; Periodontal diseases
MeSH Terms: conditions — Periodontal Diseases; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Unstimulated whole saliva samples will be collected from adult participants with periodontitis and from healthy controls. The samples will be used for electrochemical and biochemical analyses of salivary biomarkers related to inflammation, oxidative stress, and microbial activity. No DNA or genetic material will be extracted. Samples will be stored under controlled conditions until analysis is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Periodontitis Group: Adults diagnosed with periodontitis based on clinical criteria.
- Healthy Control Group: Adults with no clinical signs of periodontal disease.

SUMMARY:
This observational study aims to develop and validate a novel, AI-assisted electrochemical sensor platform for saliva-based diagnostics in periodontitis. Periodontitis is a chronic inflammatory disease affecting the gums and supporting tissues of the teeth. Despite its high global prevalence, early diagnosis remains challenging because the disease often progresses silently until irreversible damage has occurred.

Saliva offers a promising, non-invasive diagnostic medium that reflects both oral and systemic health. However, its biological complexity and variability have limited its clinical use. This project addresses these challenges by combining advanced electrochemical sensing with artificial intelligence (AI) and synthetic data generation to improve diagnostic precision and reliability.

The study involves the collection of saliva samples from adult participants with diagnosed periodontitis and from healthy controls. The samples will be analyzed using a modular sensor platform equipped with multiple electrodes that detect electrochemical signals from a wide range of salivary biomarkers. The sensor data will then be processed using machine learning models trained on both real and synthetic data to classify disease states.

The main goals are to:

Evaluate the performance of the electrochemical sensor array for saliva analysis.

Develop and validate AI-based algorithms for detecting and differentiating between healthy and diseased samples.

Generate feasibility data supporting future clinical implementation of saliva-based diagnostics for periodontitis.

This interdisciplinary project combines expertise in clinical dentistry, biomedical engineering, and computer science. It is conducted in collaboration between Linköping University and Malmö University, with patient sampling carried out at an affiliated dental clinic.

The study is expected to result in a working proof-of-concept device that enables real-time, non-invasive detection of periodontitis at the point of care. By enabling earlier diagnosis and more personalized treatment, this technology may transform periodontal care and serve as a foundation for future saliva-based diagnostics targeting other oral and systemic diseases.

DETAILED DESCRIPTION:
Background and Rationale Periodontitis is a chronic inflammatory disease that affects the supporting tissues of the teeth and is one of the most prevalent oral diseases worldwide. Despite its high prevalence, early diagnosis remains a major challenge, as current diagnostic tools rely on retrospective measures such as pocket depth, bleeding on probing, and radiographic bone loss. These indicators reflect past tissue destruction rather than current disease activity, leading to delayed diagnosis and treatment.

Saliva is an attractive diagnostic fluid for non-invasive, real-time disease monitoring because it contains a complex mixture of biomarkers that reflect both oral and systemic health. However, its biological variability, matrix effects, and susceptibility to contamination have limited its reliability as a diagnostic medium. To overcome these challenges, this project integrates electrochemical sensing with artificial intelligence (AI)-driven data interpretation and synthetic data generation to enable robust saliva-based diagnostics.

Study Objectives

The overall objective is to develop and validate an AI-assisted electrochemical sensor platform capable of detecting biochemical patterns in saliva associated with periodontitis. Specific aims are to:

Design and optimize a modular, multi-electrode sensor platform for saliva analysis.

Develop and validate AI algorithms for real-time signal interpretation and disease classification.

Generate feasibility and proof-of-concept data for future clinical implementation in dental care.

Study Design and Methods This is an observational study involving saliva sampling from adult participants diagnosed with periodontitis and healthy control subjects. Approximately 25 periodontitis patients and an expanded control group will be recruited from a collaborating dental clinic.

The electrochemical sensor platform will include multiple electrode types (carbon, gold, platinum, palladium), each selected for specific electrochemical and biochemical properties. The electrodes will detect a broad spectrum of salivary biomarkers, including metabolites related to inflammation, oxidative stress, and microbial activity. The system supports several analytical modes, such as differential pulse voltammetry (DPV), which provides high sensitivity and resolution across multiple analytes.

Collected saliva samples will first be tested under controlled laboratory conditions to establish baseline sensor responses. Selected samples will also undergo complementary analyses (e.g., H-NMR, LC-MS) for calibration and validation. Sensor signals will be processed and classified using supervised and unsupervised machine learning models, including support vector machines and random forests. Synthetic data augmentation, based on generative models such as variational autoencoders, will be used to increase dataset diversity and improve model generalization, particularly in the early phase when sample numbers are limited.

Implementation Plan The project is organized over 24 months, beginning in September 2025.

Months 1-4: Selection and benchmarking of electrode materials in artificial and healthy saliva samples.

Months 5-8: Assembly of the first prototype with integrated AI signal acquisition and secure, GDPR-compliant data transmission.

Months 9-12: Development of synthetic datasets and initial training of machine learning models.

Months 9-19: Clinical saliva sampling and iterative model refinement using new data.

Months 21-24: Real-world testing of the proof-of-concept system in a clinical setting, data analysis, and dissemination of results.

Data Handling and Analysis All collected data will be de-identified and processed according to GDPR and ethical standards. Sensor outputs will be linked to anonymized clinical metadata. Machine learning models will be evaluated based on classification accuracy, sensitivity, specificity, and robustness to biological variability. Statistical analyses will include cross-validation and performance benchmarking across electrode configurations and AI models.

Expected Outcomes and Significance The study will result in a functional proof-of-concept prototype of an AI-assisted saliva diagnostic system. The platform aims to provide rapid, non-invasive detection of periodontitis at the point of care. If successful, it will represent a paradigm shift in periodontal diagnostics, enabling earlier detection, better-targeted interventions, and improved patient outcomes.

Beyond periodontitis, the modular design of the system allows adaptation for other diseases, including oral cancer, systemic inflammation, and metabolic disorders. This flexibility enhances its long-term potential as a scalable diagnostic technology for both dental and medical applications.

Ethical Considerations and Risk Management The study has been approved by the Swedish Ethical Review Authority (reference number: 2025-04853-01). All participants will provide written informed consent prior to sample collection. The study involves minimal risk, limited to the discomfort associated with saliva sampling. No experimental treatment or invasive procedures will be performed.

Potential technical risks, such as variability in saliva samples or device performance, will be mitigated through standardized sampling protocols and iterative prototype refinement. The modular hardware design ensures that individual components can be adjusted or replaced without compromising the overall system.

Collaboration and Expertise This interdisciplinary project brings together experts in clinical dentistry, biomedical engineering, and computer science. The study is led by Assoc. Prof. Shariel Sayardoust (Linköping University and Östergötland County), with collaborators Assoc. Prof. Magnus Falk, Assoc. Prof. Julia Davies, and Dr. Erdal Akin from Malmö University. Industrial collaboration with Redoxme AB supports hardware prototyping and integration.

Together, the consortium aims to establish the foundation for next-generation saliva diagnostics that combine AI, electrochemical sensing, and patient-centered care in everyday clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Adults ≥18 years.

Able and willing to provide written informed consent.

Ability to provide an unstimulated whole saliva sample per protocol (no food, drink, gum, toothbrushing, or smoking within 60 minutes prior to sampling).

Periodontitis group: Clinical diagnosis of periodontitis according to 2018 AAP/EFP criteria (e.g., interdental CAL ≥3 mm at ≥2 non-adjacent teeth with radiographic bone loss; probing pocket depth ≥4 mm in ≥2 teeth).

Healthy control group: No clinical signs of periodontal disease (no probing depths >3 mm, bleeding on probing <10%, and no radiographic bone loss).

Exclusion Criteria:

Systemic antibiotics or systemic anti-inflammatory/immunosuppressive therapy within the past 3 months.

Periodontal therapy (scaling/root planing or surgery) within the past 6 months.

Current acute oral infection or abscess.

Systemic conditions known to markedly alter saliva composition/flow (e.g., Sjögren's syndrome, prior head-and-neck radiation, ongoing chemotherapy, uncontrolled diabetes).

Use of strongly xerogenic medications not on a stable dose ≥4 weeks, or clinically significant hyposalivation preventing sampling.

Inability to comply with sampling procedures (e.g., cannot abstain from food/drink/tobacco for 60 minutes prior to sampling).

Pregnancy or lactation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult participants (≥18 years) will be recruited from an affiliated dental clinic. The study population consists of two groups: (1) patients clinically diagnosed with periodontitis according to the 2018 AAP/EFP classification, and (2) periodontally healthy adults with no signs of periodontal disease. All participants must be able to provide informed consent and a saliva sample according to study protocol.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the AI-Assisted Electrochemical Saliva Sensor for Detecting Periodontitis | Within 24 months after study start (end of data collection and analysis).
  This outcome assesses the diagnostic accuracy of the AI-assisted electrochemical sensor platform by calculating sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and the area under the receiver operating characteristic curve (AUC). The platform analyzes electrochemical signal patterns in saliva samples, and an AI-based classification model predicts whether participants have periodontitis.
  Clinical periodontal status (periodontitis vs. periodontal health) will be established using a full-mouth clinical examination according to the 2017 World Workshop classification criteria. Diagnostic accuracy metrics from the sensor platform will be compared against this clinical gold standard.

SECONDARY OUTCOMES:
Within-Run Repeatability of Electrochemical Saliva Sensor Signals (Coefficient of Variation) | Measured throughout the 24-month study period.
  This outcome will assess the within-run repeatability of electrochemical signal measurements generated by the sensor array when analyzing saliva samples. Repeatability will be quantified using the coefficient of variation (CV%) calculated from multiple consecutive measurements of the same saliva sample under standardized laboratory conditions.
Correlation Between Sensor Outputs and Biochemical Reference Analyses | 24 month
  To evaluate the correlation between electrochemical sensor responses and conventional biochemical or molecular reference methods (e.g., LC-MS, H-NMR) for validation of analytical accuracy.
System Usability Scale (SUS) Score for Clinical Use of the AI-Assisted Saliva Sensor Platform | 24 month
  Feasibility of clinical implementation will be evaluated using the System Usability Scale (SUS), a validated 10-item questionnaire that provides a global usability score from 0 to 100. The SUS score will assess perceived usability, learnability, and integration into dental workflow among clinical staff using the AI-assisted saliva sensor platform. Higher scores indicate better usability and feasibility for routine clinical implementation.
  The SUS score will be summarized using mean and standard deviation.

IPD SHARING:
Plan to Share IPD: No